CLINICAL TRIAL: NCT06884657
Title: Propofol Level at TCI During Mannitol
Brief Title: Effect of Mannitol on Propofol Level
Acronym: level
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: mannitol; Anesthesia (Registry Identifier: Çukurova University)
Record Dates: First submitted 2025-03-03; First posted 2025-03-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-02

CONDITIONS: Mannitol Adverse Reaction
MeSH Terms: interventions — Mannitol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mannitol (Active Comparator): 2.5 ml/kg (0.5 g/kg) Mannitol will be given to all patients 15 minutes after induction and the mannitol infusion will be adjusted to be 10 minutes.
  Interventions: Drug: mannitol
- Saline (Placebo Comparator): 2.5 ml/kg saline will be given to patients 15 minutes after induction and the infusion will be adjusted to be 10 minutes.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: mannitol — 2.5 mg/kg Mannitol will be given intravenously
  Arms: Mannitol
Other: Saline — 2.5 ml/kg saline will be given as plasebo
  Arms: Saline

SUMMARY:
Group 1 will include 20 patients aged 18 years and over, American Society of Anesthesiologist (ASA) II-III class, who will undergo supratentorial tumor surgery, and Group 2 will include 20 patients who will undergo pituitary surgery without mannitol. Total intravenous anesthesia (TIVA) will be adjusted to propofol 4 µg/dl and remifentanil 2-4 µg/dl with target-controlled infusion pumps. In the mannitol group, 2.5 ml/kg (0.5 g/kg) will be given to all patients 20 minutes after induction and the mannitol infusion will be adjusted to be 10 minutes.In Group 2, mannitol will not be used and 2.5 ml/kg isotonic will be administered in 10 minutes. Both blood and urine samples will take for measurement to propofol levels.

DETAILED DESCRIPTION:
The participants will divide into the two groups. Group 1 will include 20 patients aged 18 years and over, American Society of Anesthesiologist (ASA) II-III class, who will undergo supratentorial tumor surgery, (Mannitol group) and Group 2 will include 20 patients who will undergo pituitary surgery without mannitol (Control Group). Total intravenous anesthesia (TIVA) will be adjusted to propofol 4 µg/dl and remifentanil 2-4 µg/dl with target-controlled infusion pumps. In the mannitol group, 2.5 ml/kg (0.5 g/kg) will be given to all patients 20 minutes after induction and the mannitol infusion will be adjusted to be 10 minutes.In Group 2, mannitol will not be used and 2.5 ml/kg isotonic will be administered in 10 minutes. Both blood and urine samples will take for measurement to propofol levels. Beside to standard monitoring invasive hemodynamic monitorization (cardiac output, cardiac index, stroke volume variability) and bispectral index will apply to the all participants.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) II participants
* supratentorial tumor surgery
* eligible for mannitol use
* eligible for Total intravenous anesthesia (TIVA)

Exclusion Criteria:

* American Society of Anesthesiologist (ASA) III and upper
* Chronic kidney failure
* sepsis
* multiorgan failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Serum propofol levels | Blood samples will take at intraoperatif period during total intravenous anesthesia (TIVA). (Till the 100th minutes of anesthesia)
  Blood samples will be taken during study and then propofol levels will measure at the end of study.

SECONDARY OUTCOMES:
Urine propofol levels | The sample collection will continue till the 100th minutes of anesthesia (TIVA)
  Urine samples will take during total intravenous anesthesia (TIVA). And then urine propofol levels will measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova University, Çukurova, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No